CLINICAL TRIAL: NCT06372158
Title: Effects of Liposomal Encapsulation on Calcium Powder Absorption and Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, YenPing, Lei, Assistant professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NYCU112181AE
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Other): Day 14
  Interventions: Dietary Supplement: Stage 1
- Stage 2 (Other): Day 28
  Interventions: Dietary Supplement: Stage 2

INTERVENTIONS:
Dietary Supplement: Stage 1 — Number 1-10 :General vitamin C powder group (Contains 1500 mg Ca); Number 11-20: liposomal encapsulation Ca powder group (Contains 1500 mg of Ca and lecithin and is coated)
  Arms: Stage 1
Dietary Supplement: Stage 2 — Number 11-20 :General vitamin C powder group (Contains 1500 mg Ca); Number 1-10: liposomal encapsulation Ca powder group (Contains 1500 mg of Ca and lecithin and is coated)
  Arms: Stage 2

SUMMARY:
Compared with traditional calcium supplements, liposome calcium can increase the bioavailability of calcium and reduce the waste caused by gastric acid destruction of calcium. This allows calcium to be released slowly in the intestines, reducing the risk of indigestion or other side effects caused by excessive intake at one time. Liposomal calcium can be taken orally directly. It does not need to be dissolved in water before taking like other calcium supplements, making it more convenient to use. Based on the above advantages, liposomal calcium is a relatively safe and easy-to-absorb calcium supplement, suitable for long-term use, and can meet the body's demand for calcium. According to the recommendations of the World Health Organization, the daily calcium intake for adults should be 1000-1300 mg. In Taiwan, the seventh edition of the revised reference intake of dietary nutrients for Chinese people recommends that the daily intake for adults should be 1,000 mg. The calcium dose used in this study was 500 mg. The purpose was to explore whether the sustained-release characteristics of liposome coating technology can improve the absorption rate after consuming calcium powder and achieve better bioavailability. It is expected that microlipids made by lecithin can Lipid calcium powder increases its maintenance time in the blood, thereby increasing the supplementary effect of calcium, and is an alternative to calcium supplements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-60 years old, without heart, liver, kidney, endocrine or major organic diseases (patient report), and able to fully cooperate with the experiment.

Exclusion Criteria:

1. Patients with renal insufficiency and dialysis
2. Cancer patients
3. Underweight (BMI#17) or obese (BMI#27)
4. Those taking medications for chronic diseases
5. Blood pressure systolic blood pressure # 130 mmHg or diastolic blood pressure # 85 mmHg
6. Fasting blood glucose # 100 mg/dL
7. Fasting triglycerides # 150 mg/dL, total cholesterol # 200 mg/dL
8. Have a history of vitamin C allergy
9. People suffering from mental illness
10. Pregnant and breastfeeding women
11. Patients with hemosiderosis
12. Kidney stone patients
13. Supplements for those who take calcium for a long time

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
General examination | Day 14 and 28
  BMI(Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared) and blood pressure
Hematology Test | Day 14 and 28
  Fasting blood glucose, triglycerides, total cholesterol, Blood urea nitrogen, Creatinine(Blood urea nitrogen (BUN) and creatinine tests can be used together to find the BUN-to-creatinine ratio (BUN:creatinine). A BUN-to-creatinine ratio can help your doctor check for problems, such as dehydration, that may cause abnormal BUN and creatinine levels.), GOT, GPT

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Yang Ming Chiao Tung University, Taipei, Beitou Dist.
  - National Yang Ming Chiao Tung University, Taipei

IPD SHARING:
Plan to Share IPD: No